CLINICAL TRIAL: NCT04018287
Title: Circulating miRNAs and Bone Microstructure in Adults With Hypophosphatasia
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Dr. Christian Muschitz, Ass. Prof. Dr. Christian Muschitz, Medical University of Vienna
Other Study IDs: HPP-study
Record Dates: First submitted 2019-06-13; First posted 2019-07-12 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Hypophosphatasia; Bone Diseases, Metabolic; Bone
Keywords: microRNAs, bone microstructure
MeSH Terms: conditions — Hypophosphatasia; Bone Diseases, Metabolic | interventions — MicroRNAs

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma/Serum Samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HPP-Group: 1. genetical verified hypophosphatasia
  2. age >18 years
  3. written informed consent
  4. complete serological and radiological examinations
  Interventions: Other: HR-pQCT scans, BMD measurements, bone specific circulating microRNAs (miRNAs)
- Control-Group: 1. healthy men and women without any history of musculoskeletal diseases
  2. Alkaline phosphatase (AP) in reference range
  3. written informed consent
  4. complete serological and radiological examinations
  Interventions: Other: HR-pQCT scans, BMD measurements, bone specific circulating microRNAs (miRNAs)

INTERVENTIONS:
Other: HR-pQCT scans, BMD measurements, bone specific circulating microRNAs (miRNAs) — HR-pQCT scans (XtremeCT, SCANCO Medical, Brütisellen, Switzerland) will be performed in all patients with HPP and all CTRL at the ultradistal radius and the distal tibia, using the manufacturer's standard protocol.
  Volumetric bone Mineral density (vBMD) will be carried out. The peripheral trabecular density adjacent to the cortex and the central medullary trabecular density will be automatically evaluated. Bone microstructure including trabecular bone volume fraction, trabecular number, trabecular thickness inhomogeneity of the network, cortical thickness and cortical porosity will be analyzed.
  Measurements will be carried out by two well-trained physicians and performed with the latest available software (software version 6.0). Daily crosscalibrations with standardized control phantoms (Moehrendorf, Germany) will be conducted for validation.

SUMMARY:
The aim of the study is to accomplish a complete bone status of patients with HPP using new approaches to assess bone quality.

DETAILED DESCRIPTION:
Hypophosphatasia (HPP) is a hereditary disease of bone metabolism that is not yet curable. Clinical phenotype is variable and reaches from demineralization of bone, deformation of the skeleton, microsomia and gait abnormality to breathing difficulties. Symptoms of the adult form are low-traumatic fractures, hip or thigh pain and arthropathy. Cause of the disease is a mutation in the ALPL-gene (1p36.1-p34) coding for the tissue-nonspecific isoenzyme of alkaline phosphatase (TNAP) in liver, bone and kidney. This leads to a low activity of alkaline phosphatase (AP) and elevated levels of phosphoethanolamine (PEA) in urine.

HPP is a very rare disease with a prevalence of ~1/100 000. The Medical Department II of the St. Vincent Hospital Vienna, Department of the Medical University of Vienna and the Sigmund Freud University Vienna is a department that is specialized on bone diseases and, as a member of "Orphanet", also on In particular, (i) bone microstructure as a main component of bone strength and (ii) circulating microRNAs (miRNAs) as promising biomarkers for bone diseases will be analyzed in patients with HPP and age-, and gender-matched healthy controls.

Microstructural deteriorations of cortical and trabecular bone as well as volumetric bone density (vBMD) in radius and tibia in patients with HPP will be compared to healthy individuals using HR-pQCT (High resolution peripheral quantitative computer tomography, Scanco Medical, Brütisellen). HR-pQCT is a high-resolution, non-invasive technique to measure cortical and trabecular bone mircostructures as well as vBMD at a high resolution level (82µm).

Micro-RNAs (miRNAs) are short, non-coding RNA molecules of which some have been identified as bone specific (e.g. miR-31, miR-335, miR-155, miR-29b, miR-188, miR-550a). They play a significant role in bone metabolism controlling synthesis and function of osteoblasts as well as osteoclasts.

In recent studies we could show that these microRNAs can be detected in serum and that their serum concentration correlates with the risk for osteoporotic fractures. Data for patients with HPP do not exist yet. miRNAs will be measured by qPCR (quantitative polymerase chain reaction) in serum of patients with HPP and respective controls.

In addition, measurements of areal BMD (aBMD) by DXA (Dual Energy X-ray Absorptiometry) and DXL (Dual X-ray and Laser) will be performed. Vitamin D and established bone turnover markers including PINP (N-terminal propeptide of type I collagen), CTX (collagen type 1 cross-linked C-telopeptid) and sclerostin will be analyzed. Moreover, body composition will be determined.

ELIGIBILITY:
Inclusion Criteria for Hypophosphatasia (HPP)

* genetically verified hypophosphatasia
* age >18 years
* written informed consent
* complete serological and radiological examinations

Inclusion Criteria für Controls:

* healthy men and women without any history of musculoskeletal diseases
* written informed consent
* Alkaline phosphatase (AP) in reference range
* complete serological and radiological examinations

Exclusion Criteria for both Groups:

* inflammatory diseases
* other genetic disorders affecting bone such as osteogenesis imperfecta, Ehlers-Danlos-syndrome and fibrous dysplasia
* diabetes mellitus type 1 and 2
* COPD
* chronic kidney and liver dysfunction
* systemic glucocorticoid use and glucocorticoid induced osteoporosis
* eating disorders
* HIV-infections and any malignancy including plasmacytosis and lymphoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 30 adult patients with genetical verified childhood-onset hypophophatasia. All data will be compared to a healthy, age- and gender-matched control Group (CTRL, n=30), recruited from the general population.
  Healthy controls will be matched by age and gender. All subjects will be recruited from the general population to avoid bias. The number of female and male subjects will be equal in both groups. Postmenopausal status will be taken into account.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
HR-pQCT | Assessment once after Inclusion is completed.
  non-invasively measurement of trabecular and cortical bone microstructure
microRNA pattern | Assessment once after Inclusion is completed
  bone specific circulating microRNAs (miRNAs) in the serum of adult patients

SECONDARY OUTCOMES:
DXA Scanning | Assessment once after Inclusion is completed.
  measurement of areal bone mineral density (aBMD) at the lumbar spine, radius, total body and hip by DXA • measurement of aBMD at the calcaneus by DXL
Bone Turnover Markers (BTMs) | Assessment once after Inclusion is completed.
  serological analysis of established BTMs including PINP, CTX and sclerostin

OTHER OUTCOMES:
Patient Characteristics | Assessment once after Inclusion is completed.
  Demographic and clinical Data

CONTACTS AND LOCATIONS:
Overall Officials: Roland Kocijan, Principal Investigator — Vinforce Study Group
Locations (1):
- Medical University Vienna; St. Vincent Hospital, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Haschka J, Messner Z, Feurstein J, Hadzimuratovic B, Zwerina J, Diendorfer AB, Pultar M, Hackl M, Kuzma M, Payer J, Resch H, Kocijan R. Circulating Micro-RNAs in Patients With Hypophosphatasia: Results of the First Micro-RNA Analysis in HPP. J Clin Endocrinol Metab. 2025 Sep 16;110(10):2741-2751. doi: 10.1210/clinem/dgaf080. PMID 39930630